CLINICAL TRIAL: NCT03731624
Title: The Expression Levels of Diadenosine Polyphosphates and Mucin in Mechanical Stress-related Ocular Surface Disorders
Brief Title: Diadenosine Polyphosphates and Mucin Associated With Ocular Surface Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Principal Investigator, yichensun, Principal Investigator, Assistant Professor, Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Other Study IDs: TCRD-TPE-107-07
Record Dates: First submitted 2018-10-11; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Superior Limbic Keratoconjunctivitis; Dry Eye Syndromes; Graft Vs Host Disease
MeSH Terms: conditions — Dry Eye Syndromes; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SLK
- GVHD
- Dry eye
- Control

SUMMARY:
Dry eye disease, ocular graft-versus-host disease (GVHD), and superior limbic keratoconjunctivitis (SLK) are all ocular surface disorders which mostly involve the outer surface of the eye. Many of the ocular surface disorders may result from or be aggravated by the mechanical stress from eyelid blinking. Specifically, SLK is an inflammatory ocular surface disorder characterizing by redundant superior bulbar conjunctiva. Since redundant superior bulbar conjunctiva can cause a significant mechanical force during eyelid blinking, we found that conjunctival resection with Tenon's capsule excision is helpful in relieving the symptoms of SLK patients. Therapeutic contact lens, protecting the ocular surface from the microtrauma between eyelid and ocular surface, is also an effective treatment for severe dry eye disease, ocular GVHD, and SLK. Although shearing force/mechanical stress has been studied in many different tissues and disease entities, the impact of shearing force over ocular surface is still unclear.

While the importance of mechanical stress in ocular surface disorder has been reported, the specific molecule involving the pathogenesis is still unknown. Diadenosine polyphosphates are a family of dinucleotides. They can enhance tear secretion and increase corneal wound healing rate from previous reports. Shear-stress stimuli was also noted to be able to induce diadenosine polyphosphates releasing from human corneal epithelium. In addition, mucin, one of the three components of tear film, has been greatly emphasized in the pathogenesis of dry eye disease. There are also some reports about the shearing force compensating the mucin contents in the inflammatory lung/bowel diseases. If diadenosine polyphosphates or mucin indeed play a role in mechanical stress-related ocular surface disorders, it will be a promising therapeutic targeting in the future.

DETAILED DESCRIPTION:
Ocular surface disorders are diseases involving the most outer surface of the eyeball - the transparent layers that forms the front of the eye, including cornea and conjunctiva. One of the most common ocular surface disorders is dry eye disease (DED) which has a great impact on patients' quality of life. In addition, ocular graft-versus-host disease (GVHD) and superior limbic keratoconjunctivitis (SLK) are also ocular surface disorders affecting patients' quality of life significantly.

1. Great impact of ocular surface disorders on quality of life 1.1. Impact of dry eye disease Dry eye disease (DED) is a common ocular surface disorder. Vision-related quality of life in dry eye patients is impaired and is correlated with anxiety and depression.1 Patients with DED are often evaluated by a symptom scale called ocular surface disorder index (OSDI). The OSDI is a valid and reliable scale for diagnosis and measurement of the severity of DED or other ocular surface disorder. It is also a convenient option for clinical use as a result of its shorter completion time.

   1.2. Impact of GVHD GVHD caused by alloreactive donor T cells is an important cause of nonrelapse mortality and morbidity after allogeneic hematopoietic cell transplantation (HCT). Ocular GVHD reportedly occurs in more than 50% of allogeneic HCT recipients with chronic GVHD. It can affect all parts of the eye, but the ocular surface is the most common level of involvement. Yoshi et al suggested strong correlations of serial changes in the NIH eye score, the OSDI, and the Lee eye subscale. Given that the OSDI consists of 12 items instead of the 3 for the Lee eye subscale, they found little basis for recommending the OSDI to measure change in the activity of ocular GVHD. Therefore, the Lee eye subscale might be a good choice for determining the impact of ocular GVHD on quality of life.

   1.3. Impact of SLK SLK is an ocular surface disorder characterized by unilateral or bilateral redundancy of the superior bulbar conjunctiva with inflammation of the superior tarsal and bulbar conjunctiva. There are many patients suffering by the symptoms of SLK because of its unclear etiology and no standard treatment. In addition, SLK is not easy to make a definite diagnosis, the impact of SLK on quality of life could be underestimated.
2. Mechanical stress from eyelid blinking may be an aggravating or contributing factor of ocular GVHD and SLK 2.1. The symptoms of ocular GVHD relieved by bandage soft contact lens (BSCL) application via the isolation from mechanical stress (eyelid blinking) and ocular surface The standard treatment of ocular GVHD is still not in consensus. Because of the immune reaction participating in the pathogenesis of ocular GVHD, some topical immunosuppressants, such as cyclosporine A (CsA) and tacrolimus, are applied on the patients with ocular GVHD. Allogeneic serum eye drops and autologous plasma rich in platelet-derived growth factor (PDGF) eye drops were also reported to be effective in chronic ocular GVHD patients. For medication refractory cases, punctal plugs, scleral lens, and bandage soft contact lens (BSCL) could be applied as alternative treatments for ocular GVHD patient. According to previous report, BSCL is a safe and effective treatment option that improves manifestations of ocular GVHD. BSCL can act as a barrier to further epithelial disruption and corneal nerve stimulation by the shearing force of the upper lid during the blink.

   2.2. Mechanical stress plays a role in the pathogenesis of SLK Mechanical stimulation may contribute to the pathogenesis of SLK. We speculated that this kind of physical trauma not only results in the keratinization of conjunctival epithelium, but also induced inflammatory cells and mediators, such as mast cells and cytokines, respectively. Three out of 8 SLK patients benefitted from large diameter contact lens application. Conjunctival resection with Tenon's capsule excision was also reported as a beneficial treatment for medication refractory SLK patients.
3. The expression of diadenosine polyphosphates and mucin may alter the clinical presentation or diagnosis of ocular surface disorders 3.1. Dinucleoside polyphosphates in ocular surface disorder Diadenosine polyphosphates are a family of dinucleotides, consisting of two adenosine nucleosides joined by a phosphate chain whose length can vary from 2 to 7 phosphates. They are released from nerve terminals to the extracellular milieu where they can exert actions by interacting with purinergic receptors.

   Since the levels of diadenosine tetraphosphate (Ap4A) and diadenosine pentaphosphate (Ap5A) in tears were found to be greater in all dry eye patients, these compounds could be objective markers to score dry eye. In the forced blink experiments, concentrations of the diadenosine polyphosphates rose with increasing blink frequency.13 In addition, topical application of diadenosine tetraphosphate was also noted to be able to stimulate tear secretion in vivo. Because of the higher levels of Ap4A found in refractive surgery patients during the first day after the surgery, this dinucleotide release might help in the wound healing process as well.

   3.2. Mucin in ocular surface disorder Mucin plays an important role over the ocular surface. It converts the hydrophobic corneal surface to a hydrophilic surface by adhering to the glycocalyx on the corneal microvilli. It also contributes differently to the protection of the ocular surface against allergens, pathogens, extracellular molecules, abrasive stress, and drying. MUC1 (mucin 1), 2, 4, 5AC, and 7 are the subtypes of mucin that can be found over ocular surface, including cornea, conjunctiva, goblet cell, and lacrimal gland.

   Ocular surface pathologies, i.e. dry eye syndrome or allergic conjunctivitis, are reportedly associated with alteration of expression pattern of mucin components. Although dryness of the ocular surface is a fundamental situation, local inflammation in the epithelium plays critical roles in the pathogenesis and symptom in patients with dry eye syndrome. Mucin deficiency can lead to inflammation in the ocular surface. Expression of MUC1, MUC2, MUC4, and MUC5AC are significantly lower in conjunctival epithelium gathered by impression cytology in the patients with dry eye syndrome compared with that in normal subject.18 Reduction of MUC1 expression in dry eye local tissue is reportedly most prominent and could be a marker for diagnosis or evaluation of the disease severity. Topical eye drop of Rebamipide, a drug that is capable of stimulating of mucin secretion in gastrointestinal tract or conjunctiva, is approved in Japanese government for use in the treatment of dry eye diseases.

   Mucin was also reported as an important factor contributing to some allergic keratoconjunctivitis. In the patients with atopic keratoconjunctivitis, expression of goblet cell-specific mucin, MUC5AC mRNA, was reduced and MUC16 mRNA expression was upregulated in brush cytology specimens. Besides, patients with vernal keratoconjunctivitis had increased numbers of conjunctival goblet cells from impression cytology specimen. This phenomenon also altered the levels of mucin over the ocular surface.
4. Mechanical stress can violate the levels of diadenosine polyphosphates and mucin 4.1. Diadenosine polyphosphate under mechanical stress It is known that cells under stress accumulate various dinucleoside polyphosphates, compounds suggested to function as alarmones. The release of diadenosine polyphosphates to the tears can be caused by shear stress, such as that corneal epithelial cells release these molecules as a consequence of the lid contact during the blinking process. Daily wear of rigid gas permeable lenses also can increase the levels of Ap4A due to mechanical stimulation by blinking of the corneal epithelium, and this is associated with discomfort.

4.2. Mucin under mechanical stress Gastrointestinal tract and upper airway are the organ systems filled with mucin as an important protection. MUC1 and MUC4 in the colon and MUC3 in the duodenum were upregulated in stressed animals. These findings suggest that chronic stress may affect mucin expression in the gastrointestinal tract. In addition, human bronchial epithelial cell cultures (HBECCs) are very sensitive to the mechanical stress associated with handling and pipetting. Mucin secretion at baseline in vivo occurs in a mechanically dynamic lung environment: goblet cells are exposed continuously to mechanical forces, shear stress and compressive stress, that may stimulate and/or influence the production and secretion of mucins.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* diagnosis of dry eye disease, ocular GVHD, and SLK
* patients who ever received topical medications, including artificial tears and topical steroids, at least 3 months, but refractory to the treatment
* absence of new systemic immunosuppressive medications within 1 month

Exclusion Criteria:

* pregnancy
* absolute neutrophil count less than 1000/mL
* known hypersensitivity or allergy to contact lens care products
* treatment with scleral lenses within the previous 3 months
* evidence of any active infection in the eyes
* receiving any ocular surgeries within the previous 3 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will have recruit 40 patients with ocular surface disorders (20 dry eye patients, 10 ocular GVHD patients, and 10 SLK patients) and 10 normal subjects. Tear samples and questionnaires before and after treatment (bandage soft contact lens application) will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
adenosine polyphosphate level before treatment | before treatment
  identify the levels of adenosine polyphosphate via High Performance Liquid Chromatography (HPLC) between groups
mucin level before treatment | before treatment
  identify the levels of mucin via ELISA between groups

SECONDARY OUTCOMES:
adenosine polyphosphate after treatment | post-treatment one month, three months and six months
  identify the levels of adenosine polyphosphate via HPLC between groups
mucin after treatment | post-treatment one month, three months and six months
  identify the levels of mucin via ELISA between groups

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chen Sun, MD, PhD, Principal Investigator — Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation
Locations (1):
- Taipei Tzu Chi Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No